CLINICAL TRIAL: NCT00242086
Title: Comparison of Triphasic CT, CT/PET and MR Defined Gross Tumour With Pathological Findings in Patients With Colorectal Cancer Liver Metastases
Brief Title: Comparison of Triphasic CT, PET and MR Tumour With Pathological Findings in Colorectal Cancer Liver Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-0659-C
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Liver Metastases; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: CT, PET and MRI

SUMMARY:
The purpose of this study is to correlate the MRI CT and PET appearances of colorectal liver metastases to pathologic appearance ot better understand the accuracy of imaging to determine tumor size.

DETAILED DESCRIPTION:
The purpose of this study is to correlate the MRI CT and PET appearances of colorectal liver metastases to pathologic appearance ot better understand the accuracy of imaging to determine tumor size.

ELIGIBILITY:
Inclusion Criteria:

* liver metastases from colorectal cancer undergoing liver resection

Exclusion Criteria:

* contraindication to CT, MRI or PET

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-10; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masoom Haider, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada